CLINICAL TRIAL: NCT05095220
Title: Integration and Evaluation of a Machine Learning Algorithm for Sepsis Prediction in an Electronic Health Record System - a Prospective Observational Study
Brief Title: Integration of NAVOY® Sepsis in an Electronic Health Record System
Acronym: GENIUS
Status: Completed | Type: Observational
Sponsor: AlgoDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SEP-SE-03
Record Dates: First submitted 2021-09-30; First posted 2021-10-27 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Sepsis
Keywords: sepsis; ICU; prediction; decision support; machine learning; intensive care
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort

SUMMARY:
The study aims to evaluate the performance of NAVOY® Sepsis in predicting the sepsis risk in adult ICU patients. Data collection is performed via automatic retrieval from the electronic health record system to AlgoDx proprietary cloud service where it is analysed in a simulated environment.

ELIGIBILITY:
Inclusion Criteria:

* The subject is admitted to the ICU during the enrolment period.
* The subject is 18 years of age or older at the time of admission to the ICU.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients admitted to the ICU during the enrolment period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
NAVOY® Sepsis prediction performance | 6 months
  NAVOY® Sepsis prediction output within the simulated environment will be monitored and compared to the observed fulfilment of Sepsis-3 diagnosis criteria and sepsis specific management.

SECONDARY OUTCOMES:
Integration validation | 6 months
  A technical checklist will be used in order to validate the integration between NAVOY® Sepsis and the electronic health record system.
NAVOY® Sepsis prediction results | 6 months
  The NAVOY® Sepsis predictions results indicate if the subject is at risk of developing sepsis within the coming hours. The results are not made available to ICU staff.
Fulfilment of Sepsis-3 criteria | 6 months
  The dimensions of the Sepsis-3 diagnosis criteria that the subjects meet during their ICU stay.
Sepsis specific management | 6 months
  Actions taken at the ICU specifically as part of sepsis detection, prevention, or treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Arlbrandt, MD, Principal Investigator — Southern General Hospital
Locations (1):
- Southern General Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No